CLINICAL TRIAL: NCT00791687
Title: Prenatal Corticosteroids Enhance the Antioxidant Defense System in Extremely Low Gestational Age Neonates
Brief Title: Prenatal Corticosteroids and Antioxidants in Preterm Infants
Acronym: RESOX
Status: Completed | Type: Observational
Sponsor: Fundacion Para La Investigacion Hospital La Fe (Other)
Collaborators: University of Valencia (Other); Carlos III Health Institute (Other Government)
Responsible Party: Maximo Vento, Valencian Agency for Health
Other Study IDs: PI08/0027
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Last update posted 2008-11-14 (Estimated); Status verified 2008-11

CONDITIONS: Oxidative Stress
Keywords: Antioxidant enzymes; Glutathione; Oxidative stress; Prematurity; Respiratory distress; Non enzymatic antioxidant defense system; Enzymatic antioxidant defense system
MeSH Terms: conditions — Premature Birth; Dyspnea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PRENATAL CORTICOSTEROIDS: Extremely low gestational age neonates (<28 weeks gestation) whose mothers received full course of betamethasone before delivery.
- NON PRENATAL CORTICOSTEROIDS: Extremely low gestational age neonates (<28 weeks gestation) whose mothers did not receive full course of betamethasone before delivery.

SUMMARY:
Premature infants are highly susceptible to oxidative stress because of the immaturity of their antioxidant defense system. The use of prenatal glucocorticosteroids administered to the mother improves respiratory function and overall outcome. The investigators hypothesize that prenatal glucocorticosteroids favor the expression and competence of the antioxidant defense system.

DETAILED DESCRIPTION:
This is an observational study recruiting extremely low gestational age neonates (<28 weeks gestation) whose mothers received or not full scheduled prenatal glucocorticosteroids. Healthy term newly born infants acted as controls.

At birth cord blood were drawn for the following analytical determinations: reduced and oxidized glutathione; malondialdehyde; superoxide dismutase; catalase; glutathione peroxidase; glutathione reductase; glutathione s-transferase. In addition, first urine voided was collected for ortho-tyrosine/phenylalanine and 8-hydroxy-2-oxo-deoxyguanosine/2-deoxyguanosine determination. Analytical data and clinical outcomes are compared.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age <28 weeks
* Registered used or not of prenatal glucocorticosteroids by the mother

Exclusion Criteria:

* Use of pro-or-antioxidant drugs by the mother during gestation
* Major congenital malformations
* Prenatal inflammation (E.G.:chorioamnionitis)
* Chromosomopathies
* Uncertainty about gestational age

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Extremely low gestational age neonates < 28 weeks gestation whose mothers received or not antenatal glucocorticosteroids.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2003-01; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of glutathione redox status in cord blood. | at birth

SECONDARY OUTCOMES:
Evaluation of antioxidant activity. | at birth

CONTACTS AND LOCATIONS:
Overall Officials: MAXIMO VENTO, PHD, MD, Principal Investigator — Valencian Agency of Health
Locations (1):
- Division of Neonatology; University Hospital La Fe, Valencia, Valencia, Spain

REFERENCES:
- [Background] Arima M, Kumai T, Asoh K, Takeba Y, Murano K, Goto K, Tsuzuki Y, Mizuno M, Kojima T, Kobayashi S, Koitabashi Y. Effects of antenatal dexamethasone on antioxidant enzymes and nitric oxide synthase in the rat lung. J Pharmacol Sci. 2008 Feb;106(2):242-8. doi: 10.1254/jphs.fp0060844. Epub 2008 Feb 9. PMID 18270477
- [Background] Chandrasekar I, Eis A, Konduri GG. Betamethasone attenuates oxidant stress in endothelial cells from fetal lambs with persistent pulmonary hypertension. Pediatr Res. 2008 Jan;63(1):67-72. doi: 10.1203/PDR.0b013e31815b43ee. PMID 18043518
- [Background] Asikainen TM, White CW. Antioxidant defenses in the preterm lung: role for hypoxia-inducible factors in BPD? Toxicol Appl Pharmacol. 2005 Mar 1;203(2):177-88. doi: 10.1016/j.taap.2004.07.008. PMID 15710178
- [Background] Asikainen TM, White CW. Pulmonary antioxidant defenses in the preterm newborn with respiratory distress and bronchopulmonary dysplasia in evolution: implications for antioxidant therapy. Antioxid Redox Signal. 2004 Feb;6(1):155-67. doi: 10.1089/152308604771978462. PMID 14713347